CLINICAL TRIAL: NCT06595979
Title: Comparison of Intracranial Versus Intracranial Plus Intravenous Administration of Polymyxin B for the Treatment of Intracranial Infections Due to CRGNB
Brief Title: Intraventricular Administration of Intracranial Infections Caused by （Carbapenem-resistant Gram-negative Bacilli）CRGNB
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Ningbo Medical Center Lihuili Hospital (Other Government); First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0181
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Intracranial Infections
Keywords: Polymyxin B; Intracranial Administration; Carbapenem-Resistant Gram-Negative Bacteria; Intracranial infection
MeSH Terms: interventions — Polymyxin B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biological samples, such as cerebrospinal fluid (CSF) , will be collected for analysis during the study. These samples will not be used for DNA extraction or genetic testing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intracranial Administration Group: Participants in this group will receive polymyxin B administered directly into the brain (intracranial administration) without intravenous (IV) infusion.
  Interventions: Drug: Polymyxin B
- Intracranial Administration with IV Infusion Group: Participants in this group will receive polymyxin B both intracranially and via intravenous infusion.
  Interventions: Drug: Polymyxin B

INTERVENTIONS:
Drug: Polymyxin B — Participants in this group will receive polymyxin B administered directly into the brain (intracranial administration) without intravenous (IV) infusion.

SUMMARY:
This clinical trial aims to compare two methods of administering polymyxin B for treating severe brain infections caused by carbapenem-resistant Gram-negative bacteria (CRGNB). The two methods are: 1) delivering polymyxin B directly into the brain (intracranial administration) and 2) combining this with an intravenous (IV) infusion. The goal is to determine which approach is more effective in clearing the infection, improving patient outcomes, and influencing the concentration of polymyxin B in the cerebrospinal fluid (CSF). Participants in this study will be monitored for both effectiveness and safety, with a focus on CSF polymyxin B levels, to find the best treatment strategy for these challenging infections.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, regardless of gender.
2. Patients with cerebrospinal fluid (CSF) cultures showing carbapenem-resistant Gram-negative bacteria (such as Klebsiella pneumoniae, Acinetobacter baumannii, Pseudomonas aeruginosa) and polymyxin MIC ≤ 0.5 µg/ml.
3. Diagnosed with intracranial infection and have been receiving polymyxin B treatment for at least 5 days, with an external ventricular drain (EVD) in place for continuous drainage.

Exclusion Criteria:

1. Patients with known allergy to polymyxin B or other severe allergic histories that may affect the study.
2. Pregnant women or other conditions that the investigator deems unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Withdrawal Criteria:
  1. Patient requests to withdraw from the study.
  2. Patient's cerebrospinal fluid drug concentration results do not pass quality control center approval.
Sampling Method: Probability Sample
Enrollment: 222 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
30-Day All-Cause Mortality Rate | 30 days from the start of treatment
  The proportion of participants who die from any cause within 30 days of treatment initiation. This measure will help evaluate the overall survival impact of the treatment methods.
CSF Bacterial Clearance | Baseline, 1 week, 2 weeks, and 30 days after initiation of treatment.
  The rate at which bacteria are cleared from the cerebrospinal fluid (CSF). This will be assessed through CSF cultures and laboratory tests at designated time points to determine the effectiveness of the intervention in eradicating the infection.
Clinical Cure Rate | At the end of treatment (defined as the last day of the planned treatment regimen) and 30 days post-treatment
  The proportion of participants who achieve clinical cure, defined as the resolution of symptoms and signs of infection, assessed by clinical examination and relevant diagnostic criteria at the end of the study or follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: haibin dai, Doctorate, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (3):
- China (3):
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang